CLINICAL TRIAL: NCT07088796
Title: Toric Intraocular Lens Implantation in Pediatric Aphakia (Ages 3-8 Years): A Prospective Nonrandomized Clinical Trial
Brief Title: Toric Intraocular Lens Implantation for Pediatric Aphakia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jin Yang, Professor, Eye & ENT Hospital of Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EENT No. 2013021; No. 2013021 (Other: Fudan University Eye & ENT Hospital)
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Cataract; Congenital Cataract
Keywords: astigmatism; amblyopia; toric IOL
MeSH Terms: conditions — Astigmatism; Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analysts and investigators who observed patient outcomes during follow-up were blinded to minimize bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- toric group (Experimental): Name of Intervention: Implantation of AcrySof IQ Toric Intraocular Lens (IOL) SN6AT3-T9 Manufacturer: Alcon Laboratories, Inc.
  Details of Intervention:
  The intervention involves the surgical implantation of a toric intraocular lens (IOL) in pediatric cataract patients. This specific IOL model (SN6AT3-T9) is designed to correct astigmatism.
  Interventions: Device: Toric IOL implantation
- non-toric group (Active Comparator): Name of Intervention: Implantation of AcrySof IQ Hydrophobic Acrylic Intraocular Lens (IOL) SN60WF Manufacturer: Alcon Laboratories, Inc.
  Details of Intervention:
  The control intervention involves the surgical implantation of a non-toric, hydrophobic acrylic intraocular lens (IOL) in pediatric cataract patients. This IOL model (SN60WF) provides clear vision but does not correct pre-existing corneal astigmatism.
  Interventions: Device: Non-toric IOL implantation

INTERVENTIONS:
Device: Toric IOL implantation — All surgeries were performed by the same surgeon (J.Y.) using a standardized surgical technique (phacoemulsification for cataract extraction+ IOL implantation + anterior vitrectomy) under general anesthesia. Scleral tunnel incision was created firstly. Thereafter, 5.0-5.2mm anterior capsule capsulorrhexis, and cataract aspiration were performed. A single-piece hydrophobic acrylic IOL (SN6AT3-T9) was implanted into the capsular bag. After the corneal incision was closed with 10-0 sutures, a posterior capsulectomy of 3-4 mm and anterior vitrectomy were performed through the pars plana using 25-gauge instrumentation with high cutting frequency (3,000 to 4,000 cuts per minute) and low aspiration pressure (300 to 350 mm Hg) in all eyes. A 3.5-4.0 mm posterior capsule capsulorrhexis and anterior vitrectomy were performed in patients.
  Arms: toric group
Device: Non-toric IOL implantation — All surgeries were performed by the same surgeon (J.Y.) using a standardized surgical technique (phacoemulsification for cataract extraction+ IOL implantation + anterior vitrectomy) under general anesthesia. Scleral tunnel incision was created firstly. Thereafter, 5.0-5.2mm anterior capsule capsulorrhexis, and cataract aspiration were performed. A single-piece hydrophobic acrylic IOL (SN60WF) was implanted into the capsular bag. After the corneal incision was closed with 10-0 sutures, a posterior capsulectomy of 3-4 mm and anterior vitrectomy were performed through the pars plana using 25-gauge instrumentation with high cutting frequency (3,000 to 4,000 cuts per minute) and low aspiration pressure (300 to 350 mm Hg) in all eyes. A 3.5-4.0 mm posterior capsule capsulorrhexis and anterior vitrectomy were performed in patients.
  Arms: non-toric group

SUMMARY:
Here, we conducted a nonrandomized clinical trial aims to evaluate and compare the prognosis of visual function in children of these two types of IOL implantation over a three-year postoperative period.

ELIGIBILITY:
Inclusion Criteria: 1) aged 3 to 8 years and diagnosed as pediatric cataract; 2) at least 2.0 D of regular corneal astigmatism.

-

Exclusion Criteria: 1)history of ocular comorbidities such as such as glaucoma, retinal detachment, persistent fetal vasculature, and any retina-related pathologies; 2)history of ocular trauma or surgery; 3) concurrent severe systemic diseases; 4) lack of cooperation with slit-lamp examination, pentcam, IOL master700, subjective manifest refraction and other eye examinations.

-

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2017-10-07 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
BCVA at 3 years after surgery | 3 years after surgery

SECONDARY OUTCOMES:
UDVA | Postoperative 1 week, 2 weeks, 1 month, 3 months, 6 months, 1 year, 2 years, and 3 years.
CDVA | Postoperative 1 week, 2 weeks, 1 month, 3 months, 6 months, 1 year, 2 years, and 3 years
IOP | Postoperative day 1, 1 week, 2 weeks, 1 month, 3 months, 6 months, 1 year, 2 years, and 3 years
Axial length | Postoperative 1 month, 3 months, 6 months, 1 year, 2 years, and 3 years
stereopsis | Postoperative 6 months, 1 year, 2 years, and 3 years
residual astigmatism | Postoperative 1 week, 2 weeks, 1 month, 3 months, 6 months, 1 year, 2 years, and 3 years
Corneal astigmatism | Postoperative 1month, 3 months, 6 months, 1 year, 2 years, and 3 years.
spherical equivalent | Postoperative 1 month, 3 months, 6 months, 1 year, 2 years, and 3 years.
IOL rotation | Postoperative 1 week, 2 weeks, and 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, Ph.D, Study Chair — Fudan University
Locations (1):
- Eye and ENT hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided